CLINICAL TRIAL: NCT02885103
Title: Effect of Nasal Highflow in Combination With a Nebulizer on Reversibility in Lung Function in Patients With COPD
Brief Title: Combination of NHF and Nebulizer on Lung Function in COPD
Acronym: AEROFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Responsible Party: Principal Investigator, Jens Bräunlich, MD, MD, University of Leipzig
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 349-15-24082015
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: NHF; nasal highflow
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- inhalation with nebulizer (Placebo Comparator): inhalation with an nebulizer via mouth
  Interventions: Device: Nebulizer
- inhalation with nebulizer and NHF (Active Comparator): inhalation with combination of nebulizer and nasal high flow (NHF) via nasal cavity
  Interventions: Device: Nasal high flow (NHF)

INTERVENTIONS:
Device: Nasal high flow (NHF) — NHF will be combinated with a nebulizer. Inhalation will be done on nasal cavity.
  Arms: inhalation with nebulizer and NHF
Device: Nebulizer — Inhalation will be done will Nebulizer and via mouth
  Arms: inhalation with nebulizer

SUMMARY:
This study will prove to concept of effectiveness of NHF in combination with a nebulizer on reversibility of lung function in COPD patients.

DETAILED DESCRIPTION:
Patients will inhale on day 1 with a nebulizer and on another day with combination of nebulizer an NHF in a randomised order.

ELIGIBILITY:
Inclusion Criteria:

* stable disease
* COPD

Exclusion Criteria:

* exacerbation
* right heart decompensation
* acute respiratory insufficiency
* acute disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
changes in forced expiratory volume in 1s (FEV1) | 45 minutes
  litre
changes in breath way resistance (Rtot) | 45 min

CONTACTS AND LOCATIONS:
Overall Officials: Hubert Wirtz, MD, Study Director — University of Leipzig
Locations (1):
- Department of Respiratory Medicine, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Braunlich J, Wirtz H. Oral Versus Nasal High-Flow Bronchodilator Inhalation in Chronic Obstructive Pulmonary Disease. J Aerosol Med Pulm Drug Deliv. 2018 Aug;31(4):248-254. doi: 10.1089/jamp.2017.1432. Epub 2017 Dec 20. PMID 29261402